CLINICAL TRIAL: NCT07406074
Title: DUH Innovation Units
Brief Title: Duke Virtual IntEgrated Workflow
Acronym: Duke VIEW
Status: Not yet recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00118673
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Falls Injury; Readmission Rates; CLABSI - Central Line Associated Bloodstream Infection; Catheter Associated Urinary Tract Infection; Hospital Acquired Pressure Injury; Venous Thromboembolism (VTE); Nurses; Satisfaction, Patient; Length of Stay
Keywords: Virtual Care; Nursing; Inpatient
MeSH Terms: conditions — Venous Thromboembolism; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Clinical Unit 1: All patient beds on clinical unit 1
  Interventions: Other: Co-Care
- Clinical Unit 2: All patient beds on clinical unit 2
  Interventions: Other: Co-Care
- Clinical Unit 3: All patient beds on clinical unit 3
  Interventions: Other: Co-Care
- Clinical Unit 4: All patient beds on clinical unit 4
- Clinical Unit 5: All patient beds on clinical unit 5
- Clinical Unit 6: All patient beds on clinical unit 6

INTERVENTIONS:
Other: Co-Care — Patient care delivered together with a bedside nurse and a virtual nurse
  Groups: Clinical Unit 1; Clinical Unit 2; Clinical Unit 3

SUMMARY:
This quality improvement initiative aims to evaluate the implementation, utilization, and impact of virtual care technologies and workflows being implemented at Duke University Health System (DUHS). This project is embedded within operational workflows and is designed to inform strategic decision-making and resource allocation. The evaluation will focus on key performance indicators (KPIs) relevant to hospital operations and patient outcomes, including but not limited to: Length of Stay, Readmission Rates, Patient Satisfaction Scores, and Other Quality and Safety Metrics. These KPIs will be evaluated across three clinical units at Duke University Hospital, in which virtual care technologies are being implemented. These will be compared to three control units of similar characteristics. Differences in KPIs will be examined across all units over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the hospital on one of six clinical units

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to medical surgical floors
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-02-03 (Estimated)

PRIMARY OUTCOMES:
Falls | 12 months
  Number of patient falls in a hospital room

SECONDARY OUTCOMES:
Readmission rates | 12 months
  Rate of readmission to the hospital after discharge
Central Line-Associated Bloodstream Infection | 12 months
  Number of Central Line-Associated Bloodstream Infections
Hospital acquired pressure injury | 12 months
  Number of hospital acquired pressure injuries
Venous thromboembolism | 12 months
  Number of venous thromboembolisms
Nurse Turnover | 12 months
  Rate of nurse turnover over time
Patient Satisfaction Questionnaire (PSQ-18) | 12 months
  The PSQ is an 18-item survey designed for quick assessment of patient satisfaction with healthcare. Each item is scored on a Likert scale of 1 to 5 and has a total score range of 18 to 90, where a higher score indicates greater satisfaction.
Length of Stay | 12 months
  Average length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Shaw, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Study outcome measures will be shared
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD and supporting information will be available within three years of study completion and hosted at Duke University in the Duke Research Data Repository
Access Criteria: Data will be made available publicly in accordance with the Duke Research Data Repository
URL: https://research.repository.duke.edu/